CLINICAL TRIAL: NCT01057485
Title: Node and Atrial Fibrillation Ablation for Persistent Atrial Fibrillation
Acronym: NAFAPAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastbourne General Hospital (Other)
Responsible Party: Dr AN Sulke, NHS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAFAPAFv1.3
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-01

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AF ablation and AV node ablation (Experimental): Patients will receive the combined procedure of AF ablation as well as AV node ablation
  Interventions: Procedure: AF ablation and AV node ablation
- AV node ablation (Active Comparator): Patient will receive AV node ablation alone
  Interventions: Procedure: AV node ablation

INTERVENTIONS:
Procedure: AF ablation and AV node ablation — AF ablation and AV node ablation
  Arms: AF ablation and AV node ablation
Procedure: AV node ablation — AV node ablation
  Arms: AV node ablation

SUMMARY:
The purpose of the study is to assess combining AF ablation, with AV node ablation and pacemaker implantation for patients suffering with 'irregular heartbeats' or atrial fibrillation. The study will last 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic drug refractory atrial fibrillation.
* Patients who have had pacemaker implantation and AV node ablation with ongoing symptoms.
* Patients will already be refractory to at least 2 rate or rhythm control drugs.
* Patients must be over 18 years old.
* Patients give informed consent form prior to participating in this study.

Exclusion Criteria:

* Patient is suffering with unstable angina in last 1 week.
* Patient has had a myocardial infarction within last 2 months.
* Patient is expecting or has had major cardiac surgery within last 2 months.
* Patient is participating in a conflicting study.
* Patient is unable to perform exercise testing.
* Patient is mentally incapacitated and cannot consent or comply with follow-up.
* Patient has NYHA class III/ IV heart failure.
* Patient has LVEF <35% not secondary to tachycardia.
* Pregnancy.
* Patient suffers with other cardiac rhythm disorders.
* Recent coronary artery intervention or other factors suggesting clinical instability (ECG, clinical or laboratory findings).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
To measure the two treatment effects on VO2 max over time by means of cardiopulmonary exercise testing.To measure the two treatment effects on 6-minute hall walk distance.Echocardiographic parameters | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Eastbourne District General Hospital, Eastbourne, East Sussex, United Kingdom